CLINICAL TRIAL: NCT02227745
Title: Efficacy of Dorzolamide as an Adjuvant to Improve Visual Function After Focal Photocoagulation Treatment in Diabetic Patients With Clinically Significant Macular Edema
Brief Title: Efficacy of Dorzolamide as an Adjuvant After Focal Photocoagulation in Clinically Significant Macular Edema
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Juarez de Mexico (Other Government)
Responsible Party: Principal Investigator, Virgilio Lima Gomez, PhMD, retinology, Hospital Juarez de Mexico
Other Study IDs: HJM 2296/14-R
Record Dates: First submitted 2014-08-26; First posted 2014-08-28 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Diabetic Retinopathy; Diabetic Macular Edema
MeSH Terms: conditions — Diabetic Retinopathy | interventions — dorzolamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Dorzolamide hydrochloride (2%): dorzolamide: diabetic patients with clinical significally macular edema with treatment photocoagulation dorzolamide (2%) application 1 drop every 8 hours for 4 weeks
  Interventions: Drug: Dorzolamide hydrochloride (2%)
- Placebo Sodium hyaluronate4mg: placebo: diabetic patients with clinically significant macular edema(focal), with photocoagulation sodium hyaluronate (0.5%) application 1 drop every 8 hours for 4 weeks
  Interventions: Drug: Placebo Sodium hyaluronate 4mg

INTERVENTIONS:
Drug: Dorzolamide hydrochloride (2%) — Subsequently photocoagulation treatment was applied according to the guidelines of the ETDRS, reevaluate the patient at 4 weeks.
  Patient 1 drop of topical drug in the treaty provided every 8 hours for 4 weeks eye and again 4 weeks after cited for evaluation will be placed
  Other Names: Pio-bag (2%); Iop-Sox (2%)
  Groups: Dorzolamide hydrochloride (2%)
Drug: Placebo Sodium hyaluronate 4mg — Intervention: Subsequently photocoagulation treatment was applied according to the guidelines of the ETDRS, reevaluate the patient at 4 weeks.
  Patient 1 drop of topical drug in the treaty provided every 8 hours for 4 weeks eye and again 4 weeks after cited for evaluation will be placed.
  Other Names: Zonaker (0.5%)
  Groups: Placebo Sodium hyaluronate4mg

SUMMARY:
Photocoagulation is the standard treatment in the focal EMCS, disrupts vascular leakage and allows the pigment epithelium remove the intraretinal fluid is effective in reducing the incidence of visual loss but can reduce contrast sensitivity and retinal sensitivity, the characteristics of the function can be reduced such as setting (location and stability) are relevant to the quality of the patient's vision parameters, reading comprehension, especially the ability, duration of diabetic macular edema, could have a significant impact on survival and / or the functional reserve of the macular cells subjected to mechanical and toxic stress-induced edema. It seems that in the treatment of patients with EMCS, photoreceptor damage occurs as a recent phenomenon, and can precede neurodegeneration retinal photoreceptor loss, whereby visual function can be decreased. An adjunctive treatment as Dorzolamide facilitating effect helping resorption of intraretinal fluid through EPR and reduce adverse events that is the loss of contrast sensitivity and retinal sensitivity, response time of photocoagulation treatment could be reduced to the patient, because the rate of resorption of intraretinal fluid is facilitated and thus the duration of the response, also could reduce damage to vision caused by the inadequacies of the photoreceptors during the evolution of macular edema avoiding moderate visual loss, there by increasing the quality of life in terms of improving the quality of vision in diabetic patients. In addition to obtaining a specific adjuvant treatment with photocoagulation is helpful for focal edema in diabetic and a new level using dorzolamide in retina Dorzolamide as adjunctive therapy after focal photocoagulation is more effective than placebo in improving visual function in patients with diabetic macular edema

DETAILED DESCRIPTION:
Patients referred to ophthalmology for developing type 2 diabetes subspecialist ophthalmologist evaluate the macula them by biomicroscopy, pupillary dilation, to detect clinically significant macular edema. EMCS diagnosis is made according to ETDRS criteria, and patients who were requested to submit fluorescein angiography.

Patients presenting with focal leakage on angiography were scheduled focal photocoagulation; day focal photocoagulation is measured before the procedure Measurement of visual acuity, visual acuity, refraction Measuring contrast sensitivity Measurement of retinal sensitivity Measurement of Optical Coherence Tomography ophthalmoscopic review

Subsequently photocoagulation treatment was applied according to the guidelines of the ETDRS (1-50 number of shots, shot diameter of 100 microns and 120-180 mW power) and the patient was re-evaluated at 4 weeks, which will repeat the testing day photocoagulation.

The patient what the research project will be discussed, will be invited to participate, will be read and informed consent was explained, questions and concerns will be clarified during the study, and patients who agree to enter the study will be assigned so random treatment.

Patient 1 drop of topical drug in the treaty provided every 8 hours for 4 weeks eye is placed, the drug provided will be needed for 4 weeks, plus a control sheet dose delivery will be provided and shall be referenced again in April weeks later for evaluation:

After 4 weeks of topical treatment, evaluation from 8:00 to 11 pm will be the same from the first date

ELIGIBILITY:
Inclusion Criteria:

* • Patients 40 to 70 years with diabetic retinopathy indistinct gender

  * Clinically significant macular edema
  * Focal Filtration in fluorescein angiography
  * Means optical transparent
  * Haemoglobin less than 7% (170)
  * Best-corrected visual acuity ≥ 20/200
  * Signed Informed Consent

Exclusion Criteria:

* • Presence of other retinal or optic nerve diseases

  * Presence of any other maculopathy
  * Patient diagnosed with allergy to sulfa
  * Patient with previous eye surgery four months
  * Patients with prior application of focal photocoagulation
  * Patients who use contact lenses 2 days before the application of photocoagulation
  * Presence of external eye disease, infection, inflammation at the time of evaluation
  * The presence of corneal disease present
  * Refractive errors higher than 6.00 D (sphere) -3.00 D (cylinder)
  * Study macular Fluorangiography Ischemia
  * Thickness of the central field> 300 microns

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the accessible population are type 2 diabetic patients treated with focal photocoagulation in Hospital Juarez Mexico
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
efficiency in visual function with dorzolamide after photocoagulation | two months
  Effectiveness of dorzolamide (2%) in visual function (visual acuity, contrast sensitivity, retinal sensitivity) after 2 months of photocoagulation (treatment for focal Clinically Significant Macular Edema)

CONTACTS AND LOCATIONS:
Overall Officials: Virgilio Lima Gomez, MD, PhD, Principal Investigator — Hospital Juárez de México; Dulce Mi Razo-Blanco Hernandez, MD, PhD, Study Chair — Hospital Juarez de Mexico; Surisadai Serafín Solis, Study Chair — Instituto Politecnico Nacional
Locations (1):
- Hospital Juarez de Mexico, Mexico City, Mexico City, Mexico